CLINICAL TRIAL: NCT04321720
Title: Dose-response Relationship of Mustard Flour Footbaths in Healthy Volunteers - a Blinded, Randomized, Controlled, Four-Arm Study With Crossover Design
Brief Title: Dose-response Relationship of Mustard Flour Footbaths in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SWI_12
Record Dates: First submitted 2020-03-17; First posted 2020-03-25 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Thermogenesis by Different-dosage Mustard Flour Footbaths
Keywords: Mustard flour footbaths; Dose-response relationship; Thermogenesis; Infrared thermography; Heart rate variability; Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3-g footbath (Experimental): Footbath with 3g mustard flour per liter of water
  Interventions: Other: 3-g mustard footbath
- 6-g footbath (Experimental): Footbath with 6g mustard flour per liter of water
  Interventions: Other: 6-g mustard footbath
- 12-g footbath (Experimental): Footbath with 12g mustard flour per liter of water
  Interventions: Other: 12-g mustard footbath
- Warm water footbath (Placebo Comparator): Footbath with warm water only
  Interventions: Other: Warm water only

INTERVENTIONS:
Other: 3-g mustard footbath — A ten-minute pre-intervention rest period followed by a 20-minute footbath with 12 l of warm water (40 °C) and 36 g mustard flour (3 g per l), followed by a ten-minute post-intervention rest period.
  Arms: 3-g footbath
Other: 6-g mustard footbath — A ten-minute pre-intervention rest period followed by a 20-minute footbath with 12 l of warm water (40 °C) and 72 g mustard flour (6 g per l), followed by a ten-minute post-intervention rest period.
  Arms: 6-g footbath
Other: 12-g mustard footbath — A ten-minute pre-intervention rest period followed by a 20-minute footbath with 12 l of warm water (40 °C) and 144 g mustard flour (12 g per l), followed by a ten-minute post-intervention rest period.
  Arms: 12-g footbath
Other: Warm water only — A ten-minute pre-intervention rest period followed by a 20-minute footbath with 12 l of warm water (40 °C), followed by a ten-minute post-intervention rest period.
  Arms: Warm water footbath

SUMMARY:
A study to explore whether different dosages of mustard flour in footbaths cause different effects on warmth development as well as on general well-being and the autonomic nervous system.

DETAILED DESCRIPTION:
This is a blinded, four-arm randomized controlled trial with crossover design to explore the dose-response relationship of footbaths with different dosages of mustard flour in healthy volunteers, compared to a placebo control (footbath with warm water only). The main focus is on thermogenesis and warmth distribution, as assessed by high-resolution infrared thermography and questionnaire data before, during and after the intervention. In addition, effects on the autonomic nervous system are assessed by measuring various parameters of heart rate variability and pulse wave analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Age between 18 and 55 years

Exclusion Criteria:

* Chronic skin lesions at the lower legs or feet
* Varicose veins grade 3 and grade 4 (Marshall stage classification)
* Chronic venous insufficiency
* Known intolerance or hypersensitivity to mustard preparations
* Cardiac arrhythmia
* Cardiac pacemaker
* Asthma bronchiale
* Consumption of HRV-modulating medication (especially tricyclic antidepressants, beta blockers)
* Pregnancy
* Insufficient knowledge of the german language

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
2-item warmth perception measure at the feet after the footbath | Immediately after the footbath, timepoint 2 (t2)
  Self-reported warmth perception at both feet, assessed with the "Herdecke warmth perception questionnaire" immediately after the footbath (t2). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.

SECONDARY OUTCOMES:
2-item warmth perception measure at the feet at time point 1 (t1) and time point 3 (t3) | Immediately before (time point 1, t1) and 10 minutes following the footbath (time point 3, t3).
  Self-reported warmth perception at both feet, assessed with the "Herdecke warmth perception questionnaire" immediately before (t1) and 10 minutes following the footbath (t3). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.
2-item warmth perception measure at the hands at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3).
  Self-reported warmth perception at both hands, assessed with the "Herdecke warmth perception questionnaire" immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.
2-item warmth perception measure at the head at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3)
  Self-reported warmth perception at the head, assessed with the "Herdecke warmth perception questionnaire" immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.
1-item overall warmth perception measure at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3)
  Self-reported overall warmth perception, assessed with the "Herdecke warmth perception questionnaire" immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3). The item is scored 0-4 (0 = cold; 4 = hot).
Warmth perception and skin stimulus at the feet during the footbath | Up to 20 minutes
  Self-reported perception of warmth and skin stimulus during the footbath, assessed with a dynamic warmth and skin stimulus visual analog scale (VAS), applied once per minute (0 = cold/no stimulus; 10 = very hot/very strong stimulus).
Well-being at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3) (length of footbath is up to 20 minutes)
  Self-reported well-being, assessed with the "Basler Befindlichkeits-Skala" (Basel Mood Questionnaire, BBS) immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3). (BBS: 16 items; 7-point rating scale; higher values represent a better outcome.)
Skin surface temperature at the feet at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3)
  Skin surface temperature (°C) at both feet, measured with high-resolution infrared thermography immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3)
Skin surface temperature at the lower legs at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3)
  Skin surface temperature (°C) at both lower legs, measured with high-resolution infrared thermography immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3)
Skin surface temperature at the hands at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3)
  Skin surface temperature (°C) at both hands, measured with high-resolution infrared thermography immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3)
Skin surface temperature in the face at t1, t2 and t3 | Immediately before (time point 1, t1), immediately after (time point 2, t2) and 10 minutes following the footbath (time point 3, t3) (length of footbath is up to 20 minutes)
  Skin surface temperature (°C) in the face, measured with high-resolution infrared thermography immediately before (t1), immediately after (t2) and 10 minutes following the footbath (t3)
Heart rate variability (HRV) analysis: HF | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  HF: High frequency power band (0.15-0.40 Hz) (ms2) from frequency domain analysis, obtained from ECG recordings throughout the intervention and the pre- and post-intervention rest periods (VitaGuard® 3100 monitor, getemed, Germany)
HRV analysis: LF | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  LF: Low frequency power band (0.04-0.15 Hz) (ms2) from frequency domain analysis (VitaGuard® 3100 monitor, getemed, Germany)
HRV analysis: LF/HF ratio | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  LF/HF ratio = ratio of two bands from frequency domain analysis: LF band (0.04-0.15 Hz), HF band (0.15-0.40 Hz) (VitaGuard® 3100 monitor, getemed, Germany)
HRV analysis: SDNN | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  SDNN: Standard deviation of normal to normal (NN) intervals (ms) (VitaGuard® 3100 monitor, getemed, Germany)
HRV analysis: RMSSD | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  RMSSD: Root mean square of successive differences (ms) (VitaGuard® 3100 monitor, getemed, Germany)
HRV analysis: pNN50 | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  pNN50: Percentage of successive NN intervals that differ from each other by more than 50 ms (%) (VitaGuard® 3100 monitor, getemed, Germany)
Pulse wave analysis: Pulse Transit Time | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  Pulse Transit Time (PTT, ms), obtained from pulse oximetry recordings throughout the intervention and the pre- and post-intervention rest periods (VitaGuard® 3100 monitor, getemed, Germany)
Pulse wave analysis: Reflection Index | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  Reflection Index (RI, %, percent), obtained from pulse oximetry recordings throughout the intervention and the pre- and post-intervention rest periods (VitaGuard® 3100 monitor, getemed, Germany)
Pulse wave analysis: Perfusion Index | Up to 40 minutes (continuous measurement from the beginning of the pre-intervention rest period to the end of the post-intervention rest-period)
  Perfusion Index (PI, %, percent), obtained from pulse oximetry recordings throughout the intervention and the pre- and post-intervention rest periods (VitaGuard® 3100 monitor, getemed, Germany)
Evening morning protocol: perception of warmth and stimulus at the feet | After footbath in the evening, before going to sleep; on the following morning, within 15 minutes after waking up
  Self-reported lasting effects of the footbaths at the feet, indicated on a seven-point rating scale (higher values represent a better outcome)
Evening morning protocol: skin condition | After footbath in the evening, before going to sleep; on the following morning, within 15 minutes after waking up
  Self-reported lasting effects of the footbaths on skin condition, indicated on a seven-point rating scale (higher values represent a better outcome)
Evening morning protocol: general well-being | After footbath in the evening, before going to sleep; on the following morning, within 15 minutes after waking up
  Self-reported lasting effects of the footbaths on general well-being, indicated on a seven-point rating scale (higher values represent a better outcome)
Morning protocol: sleep quality: seven-point rating scale | In the morning after the footbath, within 15 minutes after waking up
  Self-reported sleep quality during the night following the footbaths, indicated on a seven-point rating scale (higher values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, MD, Principal Investigator — ARCIM Institute Academic Research in Complementary and Integrative Medicine
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.